CLINICAL TRIAL: NCT01212042
Title: Multiplex Microarray Chip-Based Diagnosis of Respiratory Infections
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100200; 10-CC-0200
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2016-04-05

CONDITIONS: HIV
Keywords: Pneumonia; Pulmonary Pathogens; HIV; Immunocompromised Host; Respiratory Infection; Mycobacteria
MeSH Terms: conditions — Pneumonia; Respiratory Tract Infections; Mycobacterium Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Respiratory infections have a high associated morbidity and mortality, especially in immunocompromised patients. To initiate effective treatment of respiratory infections, it is essential that a rapid and thorough laboratory analysis of respiratory specimens be performed, given the wide range of pulmonary pathogens that can be detected in this population. Conventional microbiology is time-consuming and cumbersome, and the capability of local laboratories to assess specimens for rare or unusual pathogens is often limited. This study will evaluate if a newer technology can be effectively utilized in the identification of a broader range of infectious agents relative to conventional procedures.

Resequencing Pathogen Microarray (RPM) technology developed by TessArae , LLC which ceased operations in July 2014) uses a microarray chip to identify multiple pathogens in a clinical specimen. The technology has had limited clinical application, but early studies have shown its effectiveness in accurately identifying a large number of viral and bacterial organisms. In contrast to conventional microbiological procedures based on phenotypic traits (growth characteristic and enzymatic activity), this is microarray utilizes DNA sequence analysis to detect and identify the species, serotype/subtype, or strain of the infectious agent.

Aliquots of respiratory specimens (initially, specimens collected by bronchoalveolar lavage, BAL) from 200 patients at the NIH Clinical Center and the Washington Hospital Center will be analyzed using the customized microarray chip. The specimens will be collected as part of the patients routine clinical care. The results of the TessArray microarray analysis will not be available to the clinician and therefore will not have any effect on the clinical care of the patients.

The results of the microarray analysis from each site will be compared to that site s clinical laboratory results, and the data will be analyzed by site.

DETAILED DESCRIPTION:
Respiratory infections have a high associated morbidity and mortality, especially in immunocompromised patients. To initiate effective treatment of respiratory infections, it is essential that a rapid and thorough laboratory analysis of respiratory specimens be performed, given the wide range of pulmonary pathogens that can be detected in this population. Conventional microbiology is time-consuming and cumbersome, and the capability of local laboratories to assess specimens for rare or unusual pathogens is often limited. This study will evaluate if a newer technology can be effectively utilized in the identification of a broader range of infectious agents relative to conventional procedures.

Resequencing Pathogen Microarray (RPM) technology developed by TessArae , LLC which ceased operations in July 2014) uses a microarray chip to identify multiple pathogens in a clinical specimen. The technology has had limited clinical application, but early studies have shown its effectiveness in accurately identifying a large number of viral and bacterial organisms. In contrast to conventional microbiological procedures based on phenotypic traits (growth characteristic and enzymatic activity), this is microarray utilizes DNA sequence analysis to detect and identify the species, serotype/subtype, or strain of the infectious agent.

Aliquots of respiratory specimens (initially, specimens collected by bronchoalveolar lavage, BAL) from 200 patients at the NIH Clinical Center and the Washington Hospital Center will be analyzed using the customized microarray chip. The specimens will be collected as part of the patients routine clinical care. The results of the TessArray microarray analysis will not be available to the clinician and therefore will not have any effect on the clinical care of the patients.

The results of the microarray analysis from each site will be compared to that site s clinical laboratory results, and the data will be analyzed by site.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects may be included in this study if they:

1. Are 2 years of age and older.
2. Are being evaluated for a respiratory infection.
3. Are having respiratory specimens collected as part of their clinical evaluation.
4. Agree to have specimens stored for future research.

EXCLUSION CRITERIA:

Patients unable or unwilling to give informed consent will be excluded from the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2010-09-01; Study Completion 2016-04-05

PRIMARY OUTCOMES:
The sensitivity, compared to standard microbiological methods, of a customized TessArray microarray for the diagnosis of respiratory infections. | At time of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Kovacs, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Yen KT, Lee AS, Krowka MJ, Burger CD. Pulmonary complications in bone marrow transplantation: a practical approach to diagnosis and treatment. Clin Chest Med. 2004 Mar;25(1):189-201. doi: 10.1016/S0272-5231(03)00121-7. PMID 15062610
- [Background] Boyton RJ. Infectious lung complications in patients with HIV/AIDS. Curr Opin Pulm Med. 2005 May;11(3):203-7. doi: 10.1097/01.mcp.0000156992.53246.f8. PMID 15818180
- [Background] Hirschtick RE, Glassroth J, Jordan MC, Wilcosky TC, Wallace JM, Kvale PA, Markowitz N, Rosen MJ, Mangura BT, Hopewell PC. Bacterial pneumonia in persons infected with the human immunodeficiency virus. Pulmonary Complications of HIV Infection Study Group. N Engl J Med. 1995 Sep 28;333(13):845-51. doi: 10.1056/NEJM199509283331305. PMID 7651475